CLINICAL TRIAL: NCT01736228
Title: A Phase IIb Open-label Investigation of the Safety and Efficacy of DIABECELL [Immunoprotected (Alginate-Encapsulated) Porcine Islets for Xenotransplantation] in Patients With Type 1 Diabetes Mellitus
Brief Title: Open-label Investigation of the Safety and Efficacy of DIABECELL in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Living Cell Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCT/DIA-12
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2013-10

CONDITIONS: Type 1 Diabetes
Keywords: xenotransplantation; type 1 diabetes; porcine islets
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DIABECELL (Experimental): two transplants of 10,000 IEQ/kg DIABECELL (administered at least 12 weeks apart)- total of 20,000 IEQ/kg
  Interventions: Device: DIABECELL

INTERVENTIONS:
Device: DIABECELL — two transplants of 10,000 IEQ/kg DIABECELL (administered at least 12 weeks apart)- total of 20,000 IEQ/kg

SUMMARY:
The purpose of this study is to establish the efficacy and safety of xenotransplantation of DIABECELL [immunoprotected (alginate-encapsulated) porcine islets] in patients with established type 1 diabetes mellitus

DETAILED DESCRIPTION:
Intraperitoneal islet transplantation has the potential to ameliorate type 1 diabetes mellitus and avert the long-term consequences of chronic diabetes which cannot be achieved by conventional insulin treatment.

As donor human islets are not available in sufficient numbers, porcine islets are the best alternative source as they are recognised as the most physiologically compatible xenogeneic insulin-producing cells. Although the use of pig-derived cells raises the risk of xenotic infections, this can be minimised by obtaining cells from designated pathogen-free (DPF) animals bred in isolation and monitored to be free of specified pathogens. The worldwide experience to date in more than 200 patients who have received transplants of pig tissue has not demonstrated evidence of transmitted xenotic infections.

As animal-derived tissues have to be protected from immune rejection when transplanted into humans, transplants are usually accompanied by immunosuppressive therapy. However, porcine islets are preferably transplanted without the use of immunosuppressive drugs which cause significant morbidity. To protect them from immune rejection, the islets can be encapsulated in alginate microcapsules which permit the inward passage of nutrients and glucose and the outward passage of insulin. Alginate-encapsulated porcine islets transplanted without immunosuppressive drugs have survived rejection for many months in animal studies.

DIABECELL comprises neonatal porcine islets encapsulated in alginate microcapsules. DIABECELL has been safely transplanted in healthy and diabetic mice, rats, rabbits, dogs and non-human primates. Following DIABECELL transplants, the requirement for daily insulin was significantly reduced in diabetic rats and non-human primates.

The optimal dose and frequency of transplantation of the current DIABECELL preparation for the treatment of type 1 diabetes in humans can only be determined in clinical trials. The intention of this phase IIb clinical trial is to obtain at least 52 weeks safety and preliminary efficacy data in type 1 diabetic patients following transplantation of two effective doses of DIABECELL into the peritoneal cavity.

ELIGIBILITY:
Inclusion Criteria:

* Adults (males or females) in the age range 18 to 65 years
* Diagnosis of type 1 diabetes mellitus (minimum duration of 5 years) in accordance with the American Diabetes Association's criteria. Patients should have been treated continuously with insulin since diagnosis (Expert Committee on the Diagnosis and Classification of Diabetes Mellitus 2002)
* Patients with established brittle type I diabetes mellitus with a well-documented chronic history of metabolic instability who cannot achieve acceptable metabolic control (which may include treatment with the use of a continuous insulin infusion pump) without experiencing multiple episodes of hypoglycaemia, often with unawareness
* Patients with an HbA1C ≤12% prior to receiving their first xenotransplant
* Plasma C-peptide <0.3 ng/mL following a glucagon stimulation test (Scheen et al. 1996)
* If female, no childbearing capability (those who are more than two years postmenopausal or have undergone voluntary sterilisation can be considered for enrolment) or if childbearing potential, agree to the insertion of an intrauterine device (IUD) for the duration of the study
* Provision of written informed consent. Patients will be required to agree to comply with all tests and visits specified in the protocol, and they (and their partners/close contacts) will also be required to consent to long-term microbiological monitoring, which is an integral part of the study

Exclusion Criteria:

* Type 2 diabetes, defined as age of onset >30 years and/or a history of treatment with oral hypoglycaemic medications and/or insulin resistance (defined as an insulin dose requirement ≥1.2 U/kg/day)
* An HbA1C >12% prior to receipt of the first xenotransplant Body mass index (BMI) ≥28 kg/m2
* Active infection, with plasma C-reactive protein ≥10 mg/L at baseline
* Previous receipt of an organ, skin graft, or other tissue transplant from a human or animal donor
* Treatment with immunosuppressive medications for another medical condition
* Previous history of peritoneal disease or abnormal findings at baseline laparoscopy
* Previous abdominal surgery, excluding uncomplicated appendectomy, cholecystectomy or caesarean section
* History of pelvic inflammatory disease or endometriosis
* Inability to tolerate oral medications or a history of significant malabsorption
* HIV antibody and/or risk factors for HIV infection
* Positive hepatitis C antibody, positive hepatitis B surface antigen and hepatitis B core antibody
* Kidney disease, defined as serum creatinine >130 μmol/L in men and >110 μmol/L in women and/or urinary albumin >500 mg/L and/or haematuria and/or active urinary sediment or casts
* Diabetes microvascular complications defined as untreated, potentially vision-threatening proliferative or pre-proliferative retinopathy or maculopathy; painful peripheral neuropathy; autonomic neuropathy manifesting as postural hypotension; gastroparesis or diabetic enteropathy
* Serious comorbid conditions that are likely to affect participation in the study, including:

  1. Previous coronary heart disease manifesting as non-ST elevation myocardial infarction (NSTEMI), Q-wave infarction or unstable angina; coronary artery bypass graft (CABG); or percutaneous angioplasty
  2. Previous cerebrovascular disease manifesting as transient ischaemic attacks (TIAs) or stroke
  3. Peripheral vascular disease with previous amputation
  4. History of New York Heart Association (NYHA) class II, III or IV congestive heart failure (CHF) and/or chronic atrial fibrillation
  5. Chronic obstructive pulmonary disease (COPD) or asthma with previous hospitalisation for decompensation; a requirement for mechanical ventilation at any stage; or long-term treatment with oral corticosteroids
  6. Liver disease with abnormal liver function tests defined as serum bilirubin ≥20 µmol/L, and/or ALT ≥100 U/L, and/or GGT ≥100 U/L, and/or albumin <35 g/L
  7. Haematological disorders, including haemoglobin ≤110 g/L or platelet count <80 x 109/L
  8. Peptic ulcer disease and/or history of previous gastrointestinal bleeding
  9. Malignancy other than basal cell carcinoma
  10. History of epilepsy
  11. Untreated hypothyroidism
  12. Known adrenal insufficiency
* History of drug, substance or alcohol addiction
* Any factor detected from psychometric evaluation at Visit 2 pre-transplant during the screening period which may in the opinion of the Clinical Psychologist affect an individual's ability to fully participate in the study
* Any other condition that, in the opinion of the Investigator, may interfere with adherence to the study protocol, including dementia, mental illness, or a history of non-adherence to appointments or treatments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
to establish the efficacy and safety of DIABECELL | 52 weeks
  1. Restoration of sustained euglycaemia, in particular avoidance of severe hypoglycaemia, with a reduction in unaware hypoglycaemic events, without an increase in insulin dose
  2. Safety of xenotransplantation of DIABECELL [immunoprotected (alginate-encapsulated) porcine islets]

SECONDARY OUTCOMES:
Porcine β-cell function as demonstrated by measurement of porcine pro-insulin in xenotransplant recipients | 52 weeks
Improvement in the quality-of-life of xenotransplant recipients | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Adrián Abalovich, Principal Investigator — Eva Perón Hospital, San Martín,
Locations (1):
- Hospital Interzonal General de Agudos Eva Perón, San Martín, Buenos Aires, Argentina